CLINICAL TRIAL: NCT01179373
Title: Phase 2 Study of Trans Cranial Magnetic Stimulation as Additional Therapy Patients With Alzheimer's Disease
Brief Title: Deep Transcranial Magnetic Stimulation for Treatment of Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10003
Record Dates: First submitted 2010-08-08; First posted 2010-08-11 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- TMS, High Frequency (Active Comparator): High Frequency TMS with H coil to prefrontal cortex
  Interventions: Device: TMS, H coil
- TMS, Low Frequency (Active Comparator): Low Frequency TMS to Prefrontal cortex
  Interventions: Device: TMS, H coil
- Sham Stimulation (Placebo Comparator): Sham TMS with H Coil on Prefrontal Cortex
  Interventions: Device: TMS, H coil

INTERVENTIONS:
Device: TMS, H coil — TMS, H Coil, High/ Low Frequency
  Other Names: TransCranial Magnetic Stimulation

SUMMARY:
The primary objective of this trial is to assess the ability of Transcranial Magnetic Stimulation with H coil to prefrontal cortex , with an addition of cognitive brain training, to improve cognitive performance in patients with Alzheimer's disease which received drug treatment. This study is a single-center, double-blind 4 months duration trial.

DETAILED DESCRIPTION:
Primary outcome measure: ADAS-COG (time frame baseline, 2 months, 4 months) Secondary outcome measure: CGI-C,FAB, ADL, Neuropsychological computerized test(time frame baseline, 2 months, 4 months.

Estimated enrollment: 40 patients Estimated Study start Date: November 2008 Estimated Study Completion date: November 2009 Number of arms: 2

Ages: 50-85 Genders: both

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 50-85.
2. Diagnosed with Alzheimer's disease for at least one year (by the DSM-IV criteria).
3. Scored below 24 on the MMSE.
4. Received drug therapy for their disease, with each treatment having been administered at an acceptable dosage for at least 5 weeks, with either no effect or only partial response.
5. Answered in the negative to all questions in the pre-TMS treatment safety questionnaire.
6. Gave their oral and written consent to participate in the trial.

Exclusion criteria:

1. An additional neurological or psychiatric disorder.
2. Severe personality disorder.
3. Uncontrolled hypertension.
4. History of epilepsy, seizure, or heat convulsion.
5. History of epilepsy or seizure in first degree relatives.
6. History of head injury or stroke.
7. History of metal implants in the head (except dental fillings).
8. History of surgery entailing metallic implants or known history of any metallic particles in the eye, implanted cardiac pacemaker, cochlear implants, use of neurostimulators, or any medical pumps.
9. History of migraines in the last six months.
10. History of drug or alcohol abuse.
11. Inadequate communication with examiner.
12. Participation in another clinical study, either concurrent with this trial or in the 3 months preceding it.
13. Inability to sign a consent form.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2010-08 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
cognitive functioning score by ADAS-COG | 4 months

SECONDARY OUTCOMES:
Global advancement score by CGI-C | 4 months
Frontal lobe functioning score by FAB | 4 months
Daily activity score by ADL | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Merchav Clinics, Tel Aviv, Israel